CLINICAL TRIAL: NCT04485169
Title: Therapeutic Plasma Exchange for Coronavirus Disease-2019 Triggered Cytokine Release Storm; a Retrospective Propensity Matched Control Study
Brief Title: Therapeutic Plasma Exchange for Coronavirus Disease-2019 Triggered Cytokine Release Storm;
Acronym: Plex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNICEF (Other)
Collaborators: Pak Emirates Military Hospital Rawalpindi (Unknown)
Responsible Party: Principal Investigator, sultan mehmood kamran, Classified Medical specialist, UNICEF
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sultan Mehmood Kamran
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: COVID-19; Cytokine Release Syndrome
Keywords: Therapeutic Plasma exchange; Cytokine release storm; COVID-19; ARDS; Critical disease
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — Plasma Exchange

STUDY DESIGN:
Intervention Model Description: It was an interventional retrospective Propensity score matched (PSM) single centre based cohort study in Pak Emirates Military Hospital Rawalpindi (PEMH), Pakistan from 1st April to 30th June 2020. This study was carried out at the Department of Pulmonology and Critical care. PEMH is the largest Covid-19 designated hospital in the country. Data of all hospitalized patients is maintained by PEMH Covid-19 Research and evaluation cell. The study was approved by Institutional Review Board.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPE Arm (Experimental): In addition to standard care TPE was performed once daily using COBE Spectra Apheresis machine version 7 (Manufacturer TERUMO BCT, Lakewood, CO, USA INC) having continuous flow centrifugation. Venous access was achieved using an ultrasound guided double lumen catheter (Arrow - 12 FR) via femoral vein. Patient's total blood volume was calculated as per Nadler's formula. Anticoagulant acid dextrose ratio was 1:10 and flow rate 30-40 ml/minutes (Adjusted as per hemodynamic status). Patients' blood pressure, pulse, oxygen saturation was monitored throughout procedure. Duration of procedure varied from 2-4 hours and 1-1.5 times total plasma volume was removed during each procedure. Replacement fluid was fresh frozen plasma (FFP) and normal saline in 2:1 respectively. All procedures were performed in intensive care or high dependency unit by Apheresis Department of PEMH. TPE was continued till recovery
  Interventions: Procedure: Therapeutic Plasma Exchange
- NON TPE arm (No Intervention): Only supportive treatment offered including Vit C, Zinc, Vit D, famotidine, Enoxaparin and Methylprednisolone

INTERVENTIONS:
Procedure: Therapeutic Plasma Exchange — a. 1-1.5 plasma volume exchange, 2/3rd plasma should be replacing with FFP to avoid coagulopathy, adequate dieresis to prevent volume overload, 1-5 sessions in total, 1 session daily
  Arms: TPE Arm

SUMMARY:
Background:

investigators have seen recently from experience in Western countries with best health care systems that pandemics cannot be managed in hospitals. Investigators have seen ICUs crowded to capacity, healthcare workers being exposed and going to quarantine or dying after exposure to large doses of viral inoculums. Investigators recommend that institutions should register for Clinical trials and consider emergency use of TPE. In Pandemics, time is of essence to avoid mortality by intervening early with available evidence, preferably as part of clinical trial.

Scientific rationale:

Beyond supportive care, there are currently no proven treatment options for coronavirus disease (COVID-19) and related pneumonia, caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). However, literature review has shown that most common cause of death in severe SARS-COV-2 is Cytokine release syndrome and Hemophygocytic Lymphohistocytosis (HLH). In this context, Investigators seek to treat patients who are sick enough to warrant hospitalization prior to the onset of overwhelming disease including a systemic inflammatory response, sepsis, and/or Acute Respiratory Distress Syndrome (ARDS).

DETAILED DESCRIPTION:
PROTOCOL SUMMARY:

Therapeutic plasma exchange for coronavirus disease-2019 triggered cytokine release storm; a retrospective propensity matched control study

Clinical Phase: Two arms, Phase 2 Open Label

Conducted by: Department of Pulmonology and Critical Care; Pak Emirates Military Hospital.

Sample Size: 280

Study Population: Hospitalized COVID-19 patients aged ≥18 years to 80 years of with Moderate- severe-critical disease and evidence of Cytokine release storm (CRS)

Study Duration: 1st April, 2020 to 31st July 2020

Study Design: A retrospective propensity matched control trial will assess the efficacy and safety of following treatment options

1. Standard treatment including steroids
2. Therapeutic plasma exchange in addition to standard treatment

Operational Definitions

1. Moderate disease:

   COVID-19 positive case with lung infiltrates < 50% of total lung fields on Chest X-ray / peripheral ground glass opacities (GGOs) on High Resolution Computerized Tomography (HRCT)chest but no evidence of hypoxemia.
2. Severe disease:

   COVID-19 pneumonia with evidence of hypoxemia (RR > 30/minute or PaO2 on ABGs < 80mmHg or PaO2/FiO2 (PF ratio) < 300 or lung infiltrates > 50% of the lung field).
3. Critical illness:

   COVID-19 pneumonia with evidence of either respiratory failure (PaO2 < 60mmHg) or multiorgan dysfunction syndrome (MODS) measured by Sequential Organ Failure assessment (SOFA score) > 10 or septic shock (Systolic BP less than 90 or less than 40mm Hg of baseline in hypertensive or Urine output < 0.5 ml/kg/hour).Age, sex, comorbidities, date of symptoms, source of infection, type of admission SOFA score, Clinical status, vital signs including temperature, respiratory rate, oxygen saturation, oxygen requirement, Complete Blood counts (CBC) with neutrophil counts, lymphocytes count, C-reactive Proteins (CRP), chest imaging (CT or X-ray), location and status in hospital
4. Cytokine release storm (CRS):

Diagnostic criteria of Cytokine release syndrome (CRS) CRS is defined as fever of equal to or more than 100 F persisting > 48 hours in absence of documented bacterial infection and ANY of the following in the presence of moderate, severe or critical disease

1. Ferritin >1000 mcg/L and rising in last 24 hours
2. Ferritin >2000 mcg/L in patient requiring high flow oxygen or ventilation
3. Lymphopenia < 800 cells/ul or lymphocyte percentage <20% and two of the following

   1. Ferritin >700 mcg/mL and rising in the last 24 hours
   2. LDH > 300 IU (reference 140-250 IU/L) and rising in the last 24 hours
   3. D-Dimer >1000ng/mL (or >1mcg/ml) and rising in the last 24 hours
   4. CRP >70 mg/L (or >10 hsCRP) and rising in the last 24 hours, in absence of bacterial infection
   5. If any 3 of above presents on admission no need to document rise

5. Standard treatment:

As per Institutional COVID-19 Management Guidelines all patients of moderate, severe and critical COVID-19 received standard protocol of aspirin, anticoagulation, ulcer prophylaxis, awake Proning (if PaO2 < 80mmHg) and corticosteroids. All patients of CRS received Methylprednisolone 1 mg/kg irrespective of disease severity.

6. Therapeutic Plasma exchange (TPE)

Therapeutic plasma exchange: 1-1.5 plasma exchange daily (1-5 sessions) with replacement fluid Fresh frozen Plasma (FFP) (whole volume) to 70 willing patients of moderate, severe and critical disease with evidence of CRS after explaining the investigational role of this therapy. TPE will be given in addition to standard treatment to 70 patients randomly. TPE related complications to be documented

7. Recovery Recovery to be defined by de-escalation of patients condition from severe to moderate, or from moderate to mild, plus at least 2 of the following; serum Ferritin < 1000 ug/ml (and decreasing trend on two consecutive days), serum LDH normalization, C-reactive protein > 50% fold reduction (and decreasing trend in on two consecutive days),), ALC > 1000 and PT/APTT normalization.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 diagnosed by Polymerase Chain Reaction (PCR) positivity for SARS-CoV2
* CRS at presentation or developing during hospitalization
* 10-80 years age and both genders
* hospital admission
* At least 1 completed session of plasma-exchange in patients included in TPE arm
* No other novel therapy administered.

Exclusion criteria were:

* Death within 48 hours of admission
* severe septic shock at time of admission
* Congestive cardiac failure (EF<20%) (4)
* Those receiving immunotherapy, Anti-thymocyte globulin or hematopoietic stem cell transplant in recent past
* Patients of hematological or solid organ malignancies
* patients receiving other investigational drugs including Tocilizumab, Convalescent plasma, Remdesivir, or Mesenchymal stem cells.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Survival | 28 days
  Death or recovery

SECONDARY OUTCOMES:
Duration of Hospitalization | 28 days
  Duration of hospitalization in days
Timing of PCR negativity | 28 days
  Time in days to achieve viral clearance
Time to CRS resolution | 28 days
  Time in days required to settle symptoms and laboratory parameters of CRS
Complications | 28 days
  Complications secondary to use of TPE

CONTACTS AND LOCATIONS:
Overall Officials: Imran m Fazal, FCPS, Study Director — Pak Emirates Military Hospital (PEMH) Rawalpindi
Locations (1):
- Pak Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
data can be shared on demand in SPSS sheet
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data is available right now and will remain available (6 months)
Access Criteria: By email

REFERENCES:
- [Background] 6. Clinical Management Guidelines for COVID-19 Infections, Version 2 [Internet]. Nhsrc.gov.pk. 2020 [cited 1 July 2020]. Available from: http://www.nhsrc.gov.pk/SiteImage/Misc/files/Clinical-Management-nfection%20v2.pdf
- [Background] Padmanabhan A, Connelly-Smith L, Aqui N, Balogun RA, Klingel R, Meyer E, Pham HP, Schneiderman J, Witt V, Wu Y, Zantek ND, Dunbar NM, Schwartz GEJ. Guidelines on the Use of Therapeutic Apheresis in Clinical Practice - Evidence-Based Approach from the Writing Committee of the American Society for Apheresis: The Eighth Special Issue. J Clin Apher. 2019 Jun;34(3):171-354. doi: 10.1002/jca.21705. PMID 31180581
- [Background] Patel P, Nandwani V, Vanchiere J, Conrad SA, Scott LK. Use of therapeutic plasma exchange as a rescue therapy in 2009 pH1N1 influenza A--an associated respiratory failure and hemodynamic shock. Pediatr Crit Care Med. 2011 Mar;12(2):e87-9. doi: 10.1097/PCC.0b013e3181e2a569. PMID 20453703
- [Background] Busund R, Koukline V, Utrobin U, Nedashkovsky E. Plasmapheresis in severe sepsis and septic shock: a prospective, randomised, controlled trial. Intensive Care Med. 2002 Oct;28(10):1434-9. doi: 10.1007/s00134-002-1410-7. Epub 2002 Jul 23. PMID 12373468
- [Background] Keith P, Day M, Perkins L, Moyer L, Hewitt K, Wells A. A novel treatment approach to the novel coronavirus: an argument for the use of therapeutic plasma exchange for fulminant COVID-19. Crit Care. 2020 Apr 2;24(1):128. doi: 10.1186/s13054-020-2836-4. No abstract available. PMID 32241301
- [Background] Shi H, Zhou C, He P, Huang S, Duan Y, Wang X, Lin K, Zhou C, Zhang X, Zha Y. Successful treatment with plasma exchange followed by intravenous immunoglobulin in a critically ill patient with COVID-19. Int J Antimicrob Agents. 2020 Aug;56(2):105974. doi: 10.1016/j.ijantimicag.2020.105974. Epub 2020 Apr 13. PMID 32298745
- [Background] Zhang L, Zhai H, Ma S, Chen J, Gao Y. Efficacy of therapeutic plasma exchange in severe COVID-19 patients. Br J Haematol. 2020 Aug;190(4):e181-e183. doi: 10.1111/bjh.16890. Epub 2020 Jun 12. No abstract available. PMID 32453903
- [Background] Ma J, Xia P, Zhou Y, Liu Z, Zhou X, Wang J, Li T, Yan X, Chen L, Zhang S, Qin Y, Li X. Potential effect of blood purification therapy in reducing cytokine storm as a late complication of critically ill COVID-19. Clin Immunol. 2020 May;214:108408. doi: 10.1016/j.clim.2020.108408. Epub 2020 Apr 1. No abstract available. PMID 32247038
- [Result] Knaup H, Stahl K, Schmidt BMW, Idowu TO, Busch M, Wiesner O, Welte T, Haller H, Kielstein JT, Hoeper MM, David S. Early therapeutic plasma exchange in septic shock: a prospective open-label nonrandomized pilot study focusing on safety, hemodynamics, vascular barrier function, and biologic markers. Crit Care. 2018 Oct 30;22(1):285. doi: 10.1186/s13054-018-2220-9. PMID 30373638